CLINICAL TRIAL: NCT02761954
Title: Variation of Cerebral Blood Flow in Anterior Cerebral and Basilar Artery in Neonates and Infants - a Prospective Study During Planed Surgery of the Infra Umbilical Region in Combined Anaesthesia
Brief Title: Variation of Cerebral Blood Flow in Anterior Cerebral and Basilar Artery in Neonates and Infants in Genreal Anesthesia With Caudal Block
Status: Completed | Type: Observational
Sponsor: Bürgerhospital Frankfurt (Other)
Responsible Party: Principal Investigator, Ivan Erceg, Oberarzt Anästhesi-Abtl., Bürgerhospital Frankfurt
Other Study IDs: Kaudal Studie
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Anesthesia
Keywords: regional anesthesia; caudal block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
With this study we want to see how the blood flow in the anterior cerebral artery (ACA) and the basilar artery (BA) after the caudal block changes.

ELIGIBILITY:
Inclusion Criteria:

* opened big fontanella
* infraumbilical surgery

Exclusion Criteria:

* cardiac or cerebral disease
* prior operation on vertebra, heart or head/brain
* malforamtion of head or vertebra
* closed fontanella
* contraindication for caudal block (von-Willebrand-Syndrome, haemophilia,...)

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and neonates undergoing a infraumbilical surgery in general anesthesia with caudal block
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
depression of blood flow in ACA & basilar artery after caudal block | one hour

IPD SHARING:
Plan to Share IPD: No